CLINICAL TRIAL: NCT04384510
Title: Placenta Accreta Spectrum International Database (PAS-ID): Project Protocol
Brief Title: Placenta Accreta Spectrum Protocol
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sherif Abdelkarim Mohammed Shazly, MBBCh, MSc, Assiut University
Other Study IDs: PAS-ID
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta | interventions — Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with placenta accreta spectrum (PAS): This cohort presents patients who were suspected or diagnosed either antenatal or intrapartum with placenta accreta spectrum
  Interventions: Procedure: Planned Cesarean hysterectomy; Procedure: Conservative management

INTERVENTIONS:
Procedure: Planned Cesarean hysterectomy — This procedure refers to planned delivery of the fetus through Cesarean incision, leaving the placenta in situ and proceeding with hysterectomy
Procedure: Conservative management — This term describes a single or combined intervention of uterine artery ligation, internal iliac artery ligation, prophylactic balloon placement in the aorta or internal iliac artery, uterine artery embolization, compression sutures, or excision and reconstruction of uterine wall

SUMMARY:
Aim of this project is to study diagnosis and management approaches of PAS and to assess safety and efficacy of different conservative approaches compared to planned hysterectomy. We aim at improving selection process and patient counselling for women who would like to consider alternatives to hysterectomy. To achieve these objectives, creation of an international database collected by PAS-experienced centers that represent all continents would promote conduction of large studies that provide higher level of evidence on different options of management of PAS

DETAILED DESCRIPTION:
Placenta accreta spectrum (PAS) is a complex placentation disorder associated with high maternal morbidity; complications of PAS include hemorrhage, blood transfusion, multiple organ failure, and death

* The incidence of PAS has been increasing steadily in response to the increase in cesarean delivery rate
* Available evidence supports planned preterm cesarean hysterectomy with the placenta left in situ as the standard treatment of PAS

However, hysterectomy is traumatic to many women due to its operative sequences, impact on fertility, and disruption of self-image. Therefore, several conservative management options were proposed as an alternative to hysterectomy

* Although many of conservative approaches yielded satisfactory results, their implementation as a part of standard protocols has been limited
* There is primarily because evidence supporting most of these approaches is limited to case series, which is insufficient to support their safety. As a sequence, clinical trials are challenged by the lack of the margin of safety that would support ethical rationale of future studies. Availability of large multicenter studies is anticipated to provide robust evidence regarding optimal management of PAS and appropriate patient selection for conservative management

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women diagnosed with PAS, aged between 18 to 48 years.
* Women should be delivered by the corresponding center.

Exclusion Criteria:

* Inadequate follow-up
* Authorization to use anonymous patient data for research purposes.

Ages: 18 Years to 48 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Women diagnosed with placenta accreta spectrum (PAS) and managed in the recuriting hospitals between 2010 and 2020, who met study selection criteria
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Failure of conservative management of placenta accreta spectrum (PAS) | from delivery to 6 months after delivery
  Need for emergency or delayed hysterectomy following trial of conservative treatment

SECONDARY OUTCOMES:
Maternal blood loss | From delivery and up to 24 hours postpartum
  Estimation of blood loss during Cesarean section in ml
Incidence of urinary injury during intraoperative management of placenta accreta spectrum (PAS) | From delivery and up to 6 weeks postpartum
  Incidence of urinary bladder and/or ureteric injury
Admission to maternal intensive care unit (ICU) after management of placenta accreta spectrum (PAS) | From delivery and up to 6 weeks postpartum
  Admission to ICU due to maternal instability
Infectious morbidity after management of placenta accreta spectrum (PAS) | From delivery and up to 6 weeks postpartum
  Incidence of sepsis and septic shock following interventions to manage PAS

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan Faculty of Medicine, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jauniaux E, Collins S, Burton GJ. Placenta accreta spectrum: pathophysiology and evidence-based anatomy for prenatal ultrasound imaging. Am J Obstet Gynecol. 2018 Jan;218(1):75-87. doi: 10.1016/j.ajog.2017.05.067. Epub 2017 Jun 24. PMID 28599899
- [Background] Silver RM, Barbour KD. Placenta accreta spectrum: accreta, increta, and percreta. Obstet Gynecol Clin North Am. 2015 Jun;42(2):381-402. doi: 10.1016/j.ogc.2015.01.014. PMID 26002174
- [Background] Silver RM, Branch DW. Placenta Accreta Spectrum. N Engl J Med. 2018 Apr 19;378(16):1529-1536. doi: 10.1056/NEJMcp1709324. No abstract available. PMID 29669225
- [Background] Sentilhes L, Kayem G, Chandraharan E, Palacios-Jaraquemada J, Jauniaux E; FIGO Placenta Accreta Diagnosis and Management Expert Consensus Panel. FIGO consensus guidelines on placenta accreta spectrum disorders: Conservative management. Int J Gynaecol Obstet. 2018 Mar;140(3):291-298. doi: 10.1002/ijgo.12410. No abstract available. PMID 29405320
- [Background] Jauniaux E, Alfirevic Z, Bhide AG, Belfort MA, Burton GJ, Collins SL, Dornan S, Jurkovic D, Kayem G, Kingdom J, Silver R, Sentilhes L; Royal College of Obstetricians and Gynaecologists. Placenta Praevia and Placenta Accreta: Diagnosis and Management: Green-top Guideline No. 27a. BJOG. 2019 Jan;126(1):e1-e48. doi: 10.1111/1471-0528.15306. Epub 2018 Sep 27. No abstract available. PMID 30260097